CLINICAL TRIAL: NCT07064382
Title: VR-based Multi-dimensional Intervention on Cognitive Function and Well-beings
Brief Title: VR-based Multi-dimensional Intervention on Cognitive Function, With AI-agents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong University of Science and Technology (Other)
Responsible Party: Principal Investigator, GE LIN KAN, Professor, Hong Kong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MiM20250101
Record Dates: First submitted 2025-06-14; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Sleepiness; Mental Health; Alzheimer Disease
MeSH Terms: conditions — Dementia; Sleepiness; Psychological Well-Being; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: two groups, one is control (usual care), one is VR-based multi-dimensional intervention, including LLMs, AI-agent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): usual care
- VR-based intervention (Experimental): Provide VR-based multi-dimensional intervention
  Interventions: Device: VR-based multi-dimensional intervention

INTERVENTIONS:
Device: VR-based multi-dimensional intervention — VR-based multi-dimensional intervention, including LLMs, AI-agents
  Arms: VR-based intervention

SUMMARY:
Virtual Reality-based multi-dimensional intervention for cognition and well-being will be provided to older adults, with AI-agents. The digital health intervention include physical activity, gamification, cognitive trainings. Cognition, like memory, spatial function, sleepiness and mental health will be studied as outcomes.

DETAILED DESCRIPTION:
In order to study the cognitive function and well-beings, qualitative methods (like questionnaires, interviews, focus groups) and quantitative methods (like ppg, ecg, eyetracker, eeg) will be used to collect data for analysis.

ELIGIBILITY:
Inclusion Criteria:

* older adults

Exclusion Criteria:

* cannot attend physical activity like pedalling rehabilitation bike
* other health issues (assessed by health professionals)

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Spatial cognition | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  mental rotation task,higher score means stronger spatial ability
Spatial cognition | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  money road map test, higher score means stronger spatial ability
Spatial cognition | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  building memory test, higher score means stronger spatial ability
Spatial cognition | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  corsi, , higher score means stronger spatial ability
Spatial cognition | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  digit span, higher score means stronger spatial ability

SECONDARY OUTCOMES:
mental health | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  UCLA loneliness, higher score means more loneliness
mental health | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  Positive and Negative Affect Schedule , 2 subscare, one is for positive, higher score means more positive affects, one is for negative, higher score mean more negetive affects
mental health | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  The World Health Organization-Five Well-Being Index (WHO-5), higher score means better mental well-being

OTHER OUTCOMES:
Sleepiness | pre-intervention, after 4 weeks, 8 weeks, 12 weeks, 16 weeks, 3 months, 6 months, 1 year, 2 year, 3 year
  Effects on sleepiness, measured by The Pittsburgh Sleep Quality Index (PSQI)

IPD SHARING:
Plan to Share IPD: No
Personal identity and health metrics are restricted and confidentially saved.